CLINICAL TRIAL: NCT07377175
Title: A Two-Phase, Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BSY001 for Injection Following Single or Multiple Doses in Healthy Subjects.
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BSY001 After Single/Multiple Doses.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Shulan (Hangzhou) Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSY001-202401
Record Dates: First submitted 2026-01-09; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Smallpox; Cowpox; Monkeypox; Poxvirus Infection
MeSH Terms: conditions — Smallpox; Cowpox; Mpox, Monkeypox; Poxviridae Infections | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SAD Cohort 1 (Experimental): A single dose of 37.5mg BSY001 for injection or placebo administered, with 6 subjects receiving BSY001 for injection and 2 subjects receiving the placebo
  Interventions: Drug: BSY001 for Injection (37.5mg); Drug: placebo-SAD
- SAD Cohort 2 (Experimental): A single dose of 75 mg BSY001 for injection or placebo administered, with 6 subjects receiving BSY001 for injection and 2 subjects receiving the placebo
  Interventions: Drug: BSY001 for Injection (75 mg); Drug: placebo-SAD
- SAD Cohort 3 (Experimental): A single dose of 150 mg BSY001 for injection or placebo administered, with 8 subjects receiving BSY001 for injection and 2 subjects receiving the placebo
  Interventions: Drug: BSY001 for Injection (150 mg); Drug: placebo-SAD
- SAD Cohort 4 (Experimental): A single dose of 200 mg BSY001 for injection or placebo administered, with 8 subjects receiving BSY001 for injection and 2 subjects receiving the placebo
  Interventions: Drug: BSY001 for Injection (200 mg); Drug: placebo-SAD
- SAD Cohort 5 (Experimental): A single dose of 300 mg BSY001 for injection or placebo administered, with 8 subjects receiving BSY001 for injection and 2 subjects receiving the placebo
  Interventions: Drug: BSY001 for Injection (300 mg); Drug: placebo-SAD
- MAD Cohort (Experimental): Administer 200 mg of BSY001 or placebo every 12 hours for 14 consecutive days. Among them, 24 subjects will receive BSY001 for injection, and the other 6 subjects will receive placebo.
  Interventions: Drug: BSY001 for Injection; Drug: placebo-MAD

INTERVENTIONS:
Drug: BSY001 for Injection (37.5mg) — A single dose of 37.5mg BSY001 for injection.
  Arms: SAD Cohort 1
Drug: BSY001 for Injection (75 mg) — A single dose of 75 mg BSY001 for injection.
  Arms: SAD Cohort 2
Drug: BSY001 for Injection (150 mg) — A single dose of 150 mg BSY001 for injection.
  Arms: SAD Cohort 3
Drug: BSY001 for Injection (200 mg) — A single dose of 200 mg BSY001 for injection.
  Arms: SAD Cohort 4
Drug: BSY001 for Injection (300 mg) — A single dose of 300 mg BSY001 for injection.
  Arms: SAD Cohort 5
Drug: placebo-SAD — A single dose for injection.
  Arms: SAD Cohort 1; SAD Cohort 2; SAD Cohort 3; SAD Cohort 4; SAD Cohort 5
Drug: BSY001 for Injection — Administer 200 mg of BSY001 every 12 hours for 14 consecutive days.
  Arms: MAD Cohort
Drug: placebo-MAD — Administer placebo every 12 hours for 14 consecutive days.
  Arms: MAD Cohort

SUMMARY:
A Two-Phase, Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BSY001 for Injection Following Single or Multiple Doses in Healthy Subjects

DETAILED DESCRIPTION:
This study is divided into two parts: a single-dose study (BSY001-A) and a multiple-dose study (BSY001-B). Subjects for BSY001-B will be enrolled only after all subjects participating in BSY001-A have completed the pharmacokinetic (PK) tests and safety follow-ups for all dose groups, and the corresponding PK parameters and preliminary safety results have been obtained.

BSY001-A: A single ascending dose study conducted in healthy subjects. The trial includes five dose groups: 37.5, 75, 150, 200, and 300 mg, starting from the low-dose group. A total of 46 subjects are planned for enrollment. For the 37.5 mg and 75 mg dose groups, 8 subjects will be enrolled in each group, with 6 receiving BSY001 for injection and 2 receiving placebo. For the 150 mg, 200 mg, and 300 mg dose groups, 10 subjects will be enrolled in each group, including 8 receiving BSY001 for injection and 2 receiving placebo. All subjects will receive a single administration of either BSY001 for injection or placebo. PK blood samples will be collected both prior to and after the initiation of dosing. Subjects who complete PK blood sampling and safety follow-ups may be discontinued from the study. Tolerability assessment will be performed on Day 4 for each dose group, and dosing of the next dose group may commence only after the Safety Monitoring Committee (SMC) confirms safety and tolerability.

BSY001-B: A randomized, double-blind, multiple-dose pharmacokinetic study conducted in healthy subjects. A total of 30 eligible subjects will be enrolled after screening, including 24 in the treatment group and 6 in the placebo group. Subjects will receive 200 mg of BSY001 for injection or placebo, administered once every 12 hours ± 10 minutes for 14 consecutive days. During hospitalization, subjects will be under centralized management by the study center, with blood sample collection and safety assessments performed as scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study, sign the informed consent form, and agree to comply with all study requirements;
2. Aged ≥ 18 years and ≤ 50 years (based on the date of signing the informed consent form), including both males and females;
3. Body Mass Index (BMI) between 19.0 and 30.0 kg/m² (19.0 and 30.0 kg/m² inclusive); for female subjects, body weight between 45.0 and 120.0 kg (45.0 kg inclusive and 120.0 kg exclusive); for male subjects, body weight between 50.0 and 120.0 kg (50.0 kg inclusive and 120.0 kg exclusive);
4. Subjects (including their partners) voluntarily adopt effective contraceptive measures from 1 month before screening to 6 months after the last administration of the study drug, and have no plans for childbearing, sperm donation, or egg donation within the next 6 months.

Exclusion Criteria:

1. Subjects with a known allergy to Tecovirimat drugs, any excipient ingredients in this product, or subjects with an allergic diathesis (allergic to ≥ 2 types of substances);
2. Subjects with clinically significant abnormal electrocardiogram (ECG) findings or QTc prolongation as determined by the investigator (e.g., QTc interval ≥ 450 ms in males and ≥ 470 ms in females, with QTc interval calculated using the Fridericia formula);
3. Subjects with a creatinine clearance rate (Cockcroft-Gault formula) < 90 mL/min;
4. Subjects with clinically significant abnormalities in physical examination, vital signs, laboratory tests, or other auxiliary examinations as determined by the investigator;
5. Subjects with current or past history of the following clinically significant diseases as determined by the investigator, including but not limited to diseases of the cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, immune system, and nervous system (e.g., epilepsy);
6. Subjects with a current or history (within the past 3 months) of bacterial, fungal, or mycobacterial infection.;
7. Subjects with known clinically significant acute/chronic viral infections;
8. Subjects with a history of severe headache or migraine;
9. Subjects who have undergone major surgery within 6 months before drug administration, or plan to undergo surgery from the time of signing the informed consent form to 1 month after the end of the trial;
10. Subjects who have donated blood or had massive blood loss (> 450 mL) within 3 months before screening;
11. Subjects who smoked more than 5 cigarettes per day within 3 months before signing the informed consent form, or cannot refrain from using any tobacco products during the trial;
12. Subjects who consumed more than 14 units of alcohol per week within 3 months before signing the informed consent form (1 unit of alcohol ≈ 360 mL of beer, or 45 mL of spirits with 40% alcohol content, or 150 mL of wine), had a positive alcohol breath test (breath alcohol content > 0 mg/100 mL), or cannot abstain from alcohol during the trial;
13. Subjects who consumed grapefruit, grapefruit juice, chocolate, strong tea, coffee, or other beverages containing caffeine or alcohol within 72 hours before drug administration, or refuse to stop consuming the aforementioned beverages and foods during the trial;
14. Subjects who plan to engage in strenuous exercise during the trial, including contact sports or collision sports;
15. Subjects with a positive urine drug screen (for morphine, methamphetamine, ketamine, 3,4-methylenedioxymethamphetamine, or tetrahydrocannabinolic acid), or a history of drug abuse or drug use within 5 years before screening;
16. Subjects with a positive result in any of the following tests: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (IgG), hepatitis C virus core antigen, human immunodeficiency virus (HIV) antibody, or treponema pallidum-specific antibody (TP-Ab);
17. Subjects who participated in other drug clinical trials within 3 months before screening (calculated starting from the time of the last drug administration in the previous trial);
18. Subjects who took any prescription drugs, over-the-counter drugs, or traditional Chinese herbal medicines within 30 days before screening;
19. Subjects with a positive pregnancy test result;
20. Subjects who cannot tolerate venipuncture, or have a history of hematophobia (fear of blood) or trypanophobia (fear of needles);
21. Subjects who developed an acute illness or required concomitant medication from the screening phase to before the first drug administration;
22. Subjects who received a vaccine within 2 weeks before screening, or plan to receive a vaccine during the trial;
23. Subjects deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Parameters (SAD) - TEAE | 10 days
  Number and percentage of TEAE
Safety and Tolerability (SAD) - Lab tests | Day 4 and day 10 post dose
  Lab tests (complete blood count, serum biochemistry, and coagulation parameters) at baseline compared to Lab tests 4 days and 10 days post dose.
Safety and Tolerability (SAD) - Physical Examination | Day 4 and Day 10
  Physical Examination at Baseline Compared to Physical Examination 4,10 Days Post Dose
Safety and Tolerability Parameters (SAD) - Vital Signs | Day 1 pre dose; Day 1, 2, 3, 4, and 10 post dose
  Vital signs at baseline compared to Vital signs (temperature, blood pressure, pulse, breath) day 1 pre dose, day 1, 2, 3, 4, and 10 post dose
Safety and Tolerability (SAD) - Electrocardiogram | Day 1 pre dose, Day 1, 4, 10 post dose
  Electrocardiogram at Baseline Compared to Electrocardiogram day 1 pre dose, 1, 4, 10 Days Post Dose
Pharmacokinetics (MAD) - Cmax | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Maximum observed plasma drug concentration.
Pharmacokinetics (MAD) - Cmax,ss | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Steady-state peak plasma concentration
Pharmacokinetics (MAD) - Cmin,ss | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Steady-state trough plasma concentration
Pharmacokinetics (MAD) - Ctrough,ss | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Steady-state trough concentration
Pharmacokinetics (MAD) - Tmax | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Time to peak concentration
Pharmacokinetics (MAD) - Tmax,ss | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Steady-state time to peak concentration
Pharmacokinetics (MAD) - AUC0-t | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Area under the plasma concentration-time curve from time 0 to the last measurable concentration
Pharmacokinetics (MAD) - AUC0-∞ | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity
Pharmacokinetics (MAD) - AUC0-12h, AUC0-24h | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Area under the plasma concentration-time curve from 0 to 12 hours and 0 to 24 hours
Pharmacokinetics (MAD) - t½,z | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Terminal elimination half-life
Pharmacokinetics (MAD) - λz | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Terminal elimination rate constant
Pharmacokinetics (MAD) - CLz | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Clearance
Pharmacokinetics (MAD) - Vz | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Apparent volume of distribution
Pharmacokinetics (MAD) - RCmax | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Accumulation ratio based on Cmax
Pharmacokinetics (MAD) - RAUC | Day 1/14 (1st/2nd dose): Within 30 min pre-dose; 0.5, 1, 2, 4, 6 ,6.5, 8, 9, 10, 12 hours post-dose. Day 4, 6, 12, 13: Within 30 min before daily first dose. 24, 48, 72, 96, 120, 144 hours after the first dose on Day 14.
  Accumulation ratio based on AUC

SECONDARY OUTCOMES:
Pharmacokinetics (SAD) - Cmax | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Maximum observed plasma drug concentration before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
Pharmacokinetics (SAD) - Tmax | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Time to reach Cmax before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
Pharmacokinetics (SAD) - AUC0-t | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Area under the plasma concentration vs. time curve (AUC) from time 0 to the last quantifiable measurement. Samples were collected before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
Pharmacokinetics (SAD) - AUC0-∞ | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  AUC from time 0 extrapolated to infinity
Pharmacokinetics - AUC0-12h | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Area under the plasma concentration vs. time curve (AUC) from time 0 to the 12-hour time-point
Pharmacokinetics (SAD) - AUC0-24h | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Area under the plasma concentration vs. time curve (AUC) from time 0 to the 24-hour time-point
Pharmacokinetics (SAD) - t1/2 z | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Terminal elimination half-life
Pharmacokinetics (SAD) - λz | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Terminal elimination rate constant
Pharmacokinetics (SAD) - CLz | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Apparent total body clearance
Pharmacokinetics (SAD) - Vz | Before administration (within 0.5 hours); and at 0.5, 1, 2, 4, 6 (immediately post-dosing), 6.5, 8, 9, 10, 12, 16, 24, 48, and 72 hours after administration.
  Apparent volume of distribution
Safety (MAD) - TEAE | 20 days
  Number and percentage of TEAE
Safety (MAD) - Lab tests | day 2~6, day 7 and day 14, day 20.
  Lab tests (complete blood count, serum biochemistry, and coagulation parameters) at baseline compared to Lab tests at day 2~6, day 7 and day 14, day 20.
Safety (MAD) - Physical Examination | Day 20
  Physical Examination at Baseline Compared to Physical Examination at day 20
Safety (MAD) - Electrocardiogram | 1 day pre dose, day 1, 2~6, 7, 14, 20.
  Electrocardiogram at Baseline Compared to Electrocardiogram 1 day pre dose, day 1, 2~6, 7, 14, 20.
Safety (MAD) - Vital Signs | day 1 pre dose, day 1, 2~6, 7,8~13, 14, and 20
  Vital signs at baseline compared to Vital signs (temperature, blood pressure, pulse, breath) day 1 pre dose, day 1, 2~6, 7,8~13, 14, and 20

CONTACTS AND LOCATIONS:
Locations (1):
- Shulan (Hangzhou) Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No